CLINICAL TRIAL: NCT05902065
Title: Biomarkers of Rehabilitation Outcome in Patients With Parkinson's Disease: Effect of a Customized Protocol on Treadmill Training With and Without Augmented Virtual Reality Application, a Randomized Controlled Trial
Brief Title: Effect of a Progressive Treadmill Training Protocol for Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Florence (Other)
Collaborators: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Principal Investigator, Francesca Cecchi, Associate Professor, University of Florence
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VIRTREAD-PD
Record Dates: First submitted 2023-05-01; First posted 2023-06-13 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Parkinson Disease; Gait, Festinating; Fall Due to Loss of Equilibrium; Gait, Unsteady; Gait, Shuffling
Keywords: Parkinson Disease; Gait rehabilitation; Balance; Falls; Physiotherapy; Rehabilitation; Biomarkers; Raman spectroscopy; extracellular vesicles
MeSH Terms: conditions — Parkinson Disease; Gait Disorders, Neurologic

STUDY DESIGN:
Intervention Model Description: Single-center, randomized controlled, single-blind trial with no-profit purpose.
Who Masked: Outcomes Assessor
Masking Description: Outcome Assessors will be blinded regarding treatment assignment, including clinicians assessing the eligibility of patients and enrolling them in the study; the evaluators (neurologist, physiatrist, psychologist, physical therapists, engineers, laboratory staff).
  Blindness will be ensured by the modality and timing of assessments at T0, T1, and T2 that will be conducted at times other than treatment and by evaluators not involved in the treadmill training. Blinding will be removed if requested by the participant at the end of the study and in case of undesirable effects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AVR Treadmill training with C-Mill (Experimental): Participants (N=30) will undergo the AVR Treadmill training intervention with 5 AVR applications named "Nature Island", "stepping stones", "walking area": "obstacles avoidance", and "track".
  Interventions: Device: AVR Treadmill training with C-Mill
- Conventional Treadmill training with C-Mill (Active Comparator): Participants (N=30) will undergo the "Traditional Treadmill" intervention.
  Interventions: Device: Conventional Treadmill training with C-Mill

INTERVENTIONS:
Device: AVR Treadmill training with C-Mill — The protocol will include three sessions per week for 8 weeks of gait training using C-Mill with AVR applications. An anchoring system will prevent possible falls, activities will be stopped on patient request, or when a heart rate considered safe will be exceeded. The patient will be supervised by a physical therapist and asked not to use lateral bars. Treatment is planned to be progressive and will be individualized to the participant's level of performance. Progression in gait speed: at the training start, gait speed will be set at 80% of the individual's overground walking speed and weekly increased by 10%, to a maximum of 120%; progression in trial duration: at the training start the duration will be set at 25' and every two weeks increased by 5'; the maximum duration of a session will reach 45'; progression in difficulty: the protocol has 5 levels for each AVR application, and the transition among levels will be set at 80% success achievement.
  Arms: AVR Treadmill training with C-Mill
Device: Conventional Treadmill training with C-Mill — The protocol will include three sessions per week for 8 weeks of gait training using C-Mill without AVR applications, walking on the treadmill. An anchoring system will prevent possible falls, activities will be stopped on patient request, or when a heart rate considered safe will be exceeded. All sessions will be supervised by a physical therapist, who will give guidance and standardized cues on walking patterns (e.g., step length). The patient will be asked not to use the lateral bars. Treatment is planned to be progressive and will be individualized to the participant's level of performance: progression in gait speed: at the training start, gait speed will be set at 80% of the individual's overground walking speed and weekly increased by 10%, to a maximum of 120%; progression in trial duration: at the training start the duration will be set at 25' and every two weeks increased by 5'; the maximum duration of a session will reach 45'.
  Arms: Conventional Treadmill training with C-Mill

SUMMARY:
The primary objective of this single-center, no-profit, longitudinal interventional randomized controlled, single-blind trial is to compare the effects of 2 different treadmill training treatments using C-Mill: the experimental one, endowed with augmented virtual reality (AVR) applications, versus the conventional one, the standard treadmill training in PD patients with gait and or balance disturbances. The main questions the study aims to answer are 1) Is the experimental treatment more effective than the conventional one? 2) Is it possible to identify predictive and indicative biomarkers of an outcome measure of rehabilitation using extracellular vesicles (cEVs) assessed by Raman spectroscopy? Participants will be randomized into two groups: the experimental group that will receive the experimental intervention, and the control group that will receive the conventional intervention. Both groups will train three times per week for 8 weeks, the first session starting from 25 minutes (25'). The experimental and the conventional treatments are planned to be progressive and will be individualized to the participant's level of performance.

Clinical, neuropsychological, and instrumental variables will be collected at baseline (T0), at the end of the treatment (T1), and 3 months after the end of treatment (T2). At 6 months after the end of treatment (T3), a phone interview will be performed. Both within-group and between-group analyses will be conducted. Biosamples will be collected at baseline (T0) and at the end of treatment (T1).

DETAILED DESCRIPTION:
Study design: single-center, no-profit, randomized controlled single-blind trial (clinicians that assessed the effect of the interventions will be blind), with an active comparator. The study reflects the design of superiority of the experimental treatment versus the standard one. The treatment arm will be assigned by randomization. The results obtained with the 2 treatments will be compared.

The sponsor of the study is the Department of Clinical and Experimental Medicine, University of Florence, Italy; the study will be performed at "Struttura Organizzativa Dipartimentale (SOD) di Riabilitazione Generale- Istituto di Ricovero e Cura a Carattere Scientifico (IRCCS) Fondazione Don Carlo Gnocchi, Florence".

Collaborators for external services:

* Movement Analysis Laboratory at IRCCS Don Carlo Gnocchi Florence
* Laboratory of Nanomedicine and Clinical Biophotonics (LABION) at IRCCS Don Carlo Gnocchi Milan

Study start and length: study started on 6 July 2022 and will terminate on December 2023.

Study length for single participant 8 months: enrollment and baseline assessment (T0), treatment (2 months duration), end-of-treatment assessment (T1), follow-up assessment at 3 months after the end of treatment (T2), telephone interview at 6 months after the end of treatment.

Primary objective: to compare the effects of an integrated rehabilitation intervention using a new treadmill training that includes AVR applications, versus a conventional treadmill-based intervention in patients with PD (Hoehn and Yahr stage II-III) affected by walking and or balance disorders.

Secondary objective: to stratify PD patients based on their biological profile and identify predictive biomarkers and biomarkers indicative of an outcome measure of rehabilitation.

Description of the intervention. The intervention includes three sessions per week for 8 weeks. The intervention will be delivered during the "on" time of patients, every day at the same time.

The experimental and the conventional treatments are planned to be progressive and customizable to the participant's level of performance:

* progression in gait speed: gait speed is set at 80% of the individual's overground walking speed at the beginning of training, and will be weekly progressively increased to a maximum of 120%
* progression in trial duration: at the beginning of training, the duration is set at 25 minutes, including 5 slots of exercises lasting 5 minutes, with a 4-minute rest between each slot; every two weeks it will be increased by 1 minute per slot, reaching a maximal duration of 45 minutes in the last two weeks of treatment;
* progression in trial difficulty (only for the experimental group): the protocol has 5 difficulty levels for each C-Mill application, and the transition among levels is set at 80% success achievement.

Safety measures: participants will exercise wearing an anti-fall device and heart rate control; when the heart rate exceeds the safety threshold (set at 75% of HRmax, i.e., 220-age for males; 200-age for females), the treadmill speed will be lowered until the parameter is normalized.

Motek's C-Mill is a newly developed treadmill for gait and balance assessment and training that will be used for the study in both groups in a safe way (with an anti-fall device application and heart rate control). It is a treadmill sensor inclusive of a force platform. The patient is instructed to avoid using the side support bars during the training. The AVR applications of the C-Mill included in the training protocol are "nature island", "stepping stones", "walking area", "obstacles avoidance", and "tracks". These applications train balance and changes in walking speed, promote gait adaptation strategies and strategies to overcome freezing of gait, in a safe and controlled environment. Moreover, feedback to promote proper walking is provided (by physiotherapists and applications) including feedback on gait parameters such as stride symmetry, stride length, and cadence.

Visits planning and assessment timing Clinical, neuropsychological, and instrumental variables will be collected at baseline (T0), at the end of the treatment (T1), and 3 months after the end of treatment (T2). At 6 months after the end of treatment (T3) a phone interview will be performed.

All the assessments will be performed at each time point (T0, T1, T2) with some exceptions: automatic acquisition of gait parameters using C-Mill in C-Gait mode will be collected only at T1 and T2; at the end of treatment (T1), a 5-point Likert scale will also be administered to register patient satisfaction; during the phone interview at T3 only the falls questionnaire will be administered.

All visits will be planned in the "on" time of patients. Pharmacological treatments should be stable until T1.

Definition of adherence: adherence to the intervention will be considered sufficient if the patient respects the times and methods of execution of the rehabilitation treatment indicated in the intervention scheme. Missing up to 5 sessions is allowed, and lost sessions will be possibly recovered at the end of treatment. In case of discontinuation of treatment (one or more sessions missed), the treatment will be restarted with the gait speed, trial duration, and level of difficulty used in the last completed session. Participants who will miss more than 5 sessions will be considered dropouts.

Sample size. The G*Power software was used to estimate the sample size. From the literature, previous studies that aimed to evaluate the effects of treadmill training other than routine (partial weight-supported treadmill training) on patients with PD had observed a high effect size (ɳ2=0.737). In our estimate, a medium effect size (f=0.25) was conservatively chosen. Assuming a statistical power of 95% and an α=0.05, the resulting sample is 22 subjects per arm. To compensate for possible drop-outs, estimated at around 35%, the enrollment of a further 16 patients is appropriate, 8 per treatment arm, reaching an estimate of 30 subjects per group.

Data analysis. For all data, the distribution will be assessed using the Kolmogorov-Smirnov test (assuming the presence of normal distribution when p>0.05). Data will then be summarised as mean and standard deviation, median and interquartile range, or absolute and percentage frequency, as appropriate. The two groups will be compared at baseline to explore significant differences in clinical and demographic variables. Both within- and between-groups analysis will be conducted to assess the effects of the treatments delivered, for both primary and secondary outcome measures. Specifically, a repeated measures ANOVA will be used with a within-factor (Time of assessment) and a between-factor (Group). Statistical analysis will be conducted using the software International Business Machines Corporation (IBM) Statistical Package for the Social Sciences (SPSS) v28.

The acquired Raman spectra will be analyzed by multivariate Principal Component Analysis - Linear Discriminant Analysis (PCA-LDA) classification. PCA will reduce the number of variables into principal components, which will be used to build the LDA model. The model will be built to discriminate clinical improvement detected as quantifiable change on clinical scales, defined based on the minimum clinically important difference, when available from the literature. Sensitivity, specificity and accuracy of the predicting model based on spectra data will be assessed. In addition, correlation analysis will be conducted to evaluate the association between spectral data and change on clinical scales recorded between the beginning and the end of the treatment. Statistical analysis of the Raman data will be performed using Origin2021 software.

Univariate analysis models will be applied to select the best prognostic markers of clinical improvement to be included in the multivariate model. For all analyses, statistical significance will be set at p<0.05

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinson's disease according to the diagnostic (POSTUMA criteria)
* Hoehn and Yahr Stage II-III
* Age>18 years
* One fall in the past 3 months/presence of postural instability /gait disturbance
* Able to walk for at least 5 minutes without assistance
* Stable drug therapy by at least 1 month
* Willingness to participate in the study, ability to understand and willingness to sign informed consent

Exclusion Criteria:

* Other pathology concurrent with gait disturbance (symptomatic arthritis involving hip/knee/ankle, stroke outcomes, severe polyneuropathy)
* Cognitive impairment capable of interfering with rehabilitation procedures, estimated as a score less than 18.58 at the Montreal Cognitive Assessment (MoCA), row score corrected according to Aiello et al, 2022
* Hallucinations
* Psychiatric disorder not controlled by current drug therapy
* Alcohol/drug use
* Uncompensated visual/auditory deficit that limits enjoyment of the cues provided by the AVR
* Communication deficit from any cause that impairs understanding of the task and the objectives of the intervention
* Recurrent episodes of severe orthostatic hypotension
* Severe cardiovascular diseases
* Patient undergoing other experimental protocol (patients regularly undergoing physical activity or sport will not be excluded)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-07-06 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean change in gait and balance parameters assessed by the Performance Oriented Mobility Assessment - POMA scale (intra-group and between-group comparisons) | T0 (baseline); T1 (end of the treatment - 8 weeks); T2 (3 months after the end of treatment)
  The POMA scale is an easily administered task-oriented test that measures an older adult's balance (9 items) and gait (7 items) abilities. Items are scored with a three-point (0-2) or a two points (0-1) scale, where "0" indicates the highest level of impairment and "2" - "1" for dichotomic items - the individual's independence. Total Balance Score = 16; Total Gait Score = 12.
Mean change in motors parameters assessed by the Modified Unified Parkinson's Disease Rating Scale (MDS-UPDRS), part III (intra-group and between-group comparisons) | T0 (baseline); T1 (end of the treatment - 8 weeks); T2 (3 months after the end of treatment)
  The MDS-UPDRS part III includes 18 items concerning the motor examination in PD, evaluating different aspects: walking, balance, speech, bradykinesia, tremor, and rigidity. Each item is scored on a five-point ordinal rating scale, ranging from 0 to 4, where "0" indicates normal function and "4" is the highest level of impairment. Some items inclusive of evaluation of a symptom in different parts of the body, e.g on the right side, on the left side, upper and lower limbs). Score range 0-132.

SECONDARY OUTCOMES:
Correlation between Raman spectra of blood cEVs and primary outcomes after patient stratification | T0 (baseline); T1 (end of the treatment - 8 weeks)
  The biological characterization of patients at T0 analyzing cEVs performed by Raman Spectroscopy will provide numerical scores that will be correlated with motor parameters obtained at T1 to identify predictive biomarkers of an outcome measure of rehabilitation
Changes in individual Raman spectra of blood-derived cEVs before and after treatment | T0 (baseline); T1 (end of the treatment - 8 weeks)
  The Raman spectrum of blood-derived cEVs before and after treatment will be compared to identify spectral differences and to monitor the effect of rehabilitation on the spectral biomarker. Changes in the presence/absence of peaks and peaks intensity will be evaluated.

OTHER OUTCOMES:
Mean changes in walking speed (intra-group and between-group comparisons). | T0 (baseline); T1 (end of the treatment - 8 weeks); T2 (3 months after the end of treatment)
  Gait speed (m/s) will be measured at both comfortable and maximum speeds using the Optogait system (http://www.optogait.com/Gait-Phases).
Mean changes in step length during walking (intra-group and between-group comparisons). | T1 (end of treatment-8 weeks); T2 (3 months after the end of treatment)
  Right and left step length (m) will be measured at both comfortable and maximum speeds using the Optogait system (http://www.optogait.com/Gait-Phases).
Mean change in walking endurance assessed with the 6-Minutes Walking Test (6MWT) (intra-group and between-group comparisons). | T0 (baseline); T1 (end of the treatment - 8 weeks); T2 (3 months after the end of treatment)
  The distance (m) walked in 6 minutes on a 30 meters walkway will be measured, indicating the greater distance, a better score
Mean change in gait adaptability assessed by C-Gait application of C-Mill (intra-group and between-group comparisons) | T1 (end of treatment - 8 weeks); T2 (3 months after the end of treatment)
  Walking-adaptability task performance was defined as the percentage of correctly performed steps relative to the projected visual objects in 6 different tasks.
  C-gait score for each task: Level×2×Performance (%) / 100. The overall assessment score was an average score based on average performance over the six walking-adaptability tasks at the higher level of difficulty, ranging from 0 (poor performance) to 8 (excellent performance).
Mean change in freezing during walking assessed by the Freezing Of Gait Questionnaire (FOG-Q) (intra-group and between-group comparisons). | T0 (baseline); T1 (end of the treatment - 8 weeks); T2 (3 months after the end of treatment)
  The FOG-Q includes 6 items that inquires about the subject's experiences of freezing during the previous week. Each item use a five-points ordinal scale, ranging from "0" (= absence of symptoms) to "4" (= more severe disturbance). Total score ranges from 0 to 24, and higher scores correspond to more severe freezing.
Mean change in postural stability (intra-group and between-group comparisons) | T0 (baseline); T1 (end of the treatment - 8 weeks); T2 (3 months after the end of treatment)
  Postural sway assessed with a dynamometric footplate (postural sway in quiet standing with opened/closed eyes).
  Lower postural sway corresponds to better stability.
Mean change in global cognitive functions assessed by the Montreal Cognitive Assessment (MoCA) (intra-group and between-group comparisons) | T0 (baseline); T1 (end of the treatment - 8 weeks); T2 (3 months after the end of treatment)
  The MoCA test is used to assess global cognitive functions. A score superior to 18.58 is required for inclusion in the study (Aiello et al, 2021); parallel versions will be administered at different time points (Siciliano et al, 2019). Higher values correspond to better cognition, range of score 0-30.
Mean change in global cognitive functions assessed by the Parkinson's disease-cognitive rating scale, italian version (PD-CRS) (intra-group and between-group comparisons) | T0 (baseline); T1 (end of the treatment - 8 weeks); T2 (3 months after the end of treatment)
  The PD-CRS is a suitable tool to assess cognition in PD, it evaluates different domains and permits to obtain a cortical and a subcortical score:
  sum of results in item 1,3,4,5,7,8,9 (range of score 0-104), represents the subcortical score; sum of results in item 2 and 6 (range of score 0-30), represents the cortical score.
  Higher scores correspond to better cognition
Mean change in attention skills assessed by Trail Making Test A and B (TMTA and TMTB) (intra-group and between-group comparisons) | T0 (baseline); T1 (end of the treatment - 8 weeks); T2 (3 months after the end of treatment)
  TMTA evaluates sustained attention and the visual search capacity, and TMTB evaluates divided attention.
  For both tests A and B time and errors will be registered. Slowness and more errors are indicative of lower performances (No range of score).
Mean change in executive functions as assessed by the Stroop Test (intra-group and between-group comparisons) | T0 (baseline); T1 (end of the treatment - 8 weeks); T2 (3 months after the end of treatment)
  The Stroop test is used to assess executive functions (time and error interference effect).
  Slowness and higher interference effect indicative of lower performances. (No range of score).
Mean change in executive functions as assessed by the Symbol Digit oral version (intra-group and between-group comparisons) | T0 (baseline); T1 (end of the treatment - 8 weeks); T2 (3 months after the end of treatment)
  Digit symbol is used for the assessment of attention and working memory. Range of score 0-110. Higher score indicative of better performance
Mean change in functional mobility assessed by the Modified Parkinson Activity Scale (MPAS) (intra-group and between-group comparisons) | T0 (baseline); T1 (end of the treatment - 8 weeks); T2 (3 months after the end of treatment)
  The MPAS scale evaluates motor skills in activities of daily living. Range of score 0-56; higher score indicative of better functional mobility.
Mean change in functional mobility assessed by the Timed up and go test (TUG) (intra-group and between-group comparisons) | T0 (baseline); T1 (end of the treatment - 8 weeks); T2 (3 months after the end of treatment)
  The TUG is a general physical performance test used to assess mobility, balance, and gait during walking, turning, and sit-to-stand tasks.
  Time is recorded during the test; less time indicative of better performances (no range of score).
Mean change in functional autonomy assessed by the modified Barthel Index (mBI) (intra-group and between-group comparisons) | T0 (baseline); T1 (end of the treatment - 8 weeks); T2 (3 months after the end of treatment)
  mBI is a scale for assessing functional independence in daily life. Range of score 0-100. Lower score corresponds to less independence.
Mean change in the quality of life assessed by the Parkinson's Disease Questionnaire Italian version (PDQ-39-IT) (intra-group and between-group comparisons) | T0 (baseline); T1 (end of the treatment - 8 weeks); T2 (3 months after the end of treatment)
  PDQ-39 is a self-report questionnaire for assessing the quality of daily life in PD. It includes 39 items assessing how often persons experience difficulty across 8 quality of life dimensions. Each item is scored on a five-point ordinal scale from 0 (=never) to 4 (always). Each dimension total score ranges from 0 (never have difficulty) to 100 (always have difficulty). The summary total score is calculated as the mean of the 8 dimension total scores. A higher score corresponds to a lower quality of life.
Mean change in the fear to fall assessed by the Falls efficacy scale, Italian version (FES-I) (intra-group and between-group comparisons) | T0 (baseline); T1 (end of the treatment - 8 weeks); T2 (3 months after the end of treatment)
  FES-I is used for the assessment of the fear-of-fall. It includes 16 items rated on a four-point scale from 1 (not confident at all) to 4 (completely confident). Total score ranges from minimum 16 (no concern about falling) to maximum 64 (severe concern about falling).
Mean change in mood assessed by the Beck Depression Inventory II, italian version (BDI) (intra-group and between-group comparisons) | T0 (baseline); T1 (end of the treatment - 8 weeks); T2 (3 months after the end of treatment)
  BDI II is used for the assessment of mood and consists of 21 items, each of whom corresponding to a symptom of depression. Each item is scored on a scale of 0-3 in a list of four statements arranged in increasing severity. Total score ranges from 0 to 63; higher scores indicates more severe depression.
Mean change in pain perception assessed by the Numerical rating scale (NRS) (intra-group and between-group comparisons) | T0 (baseline); T1 (end of the treatment - 8 weeks); T2 (3 months after the end of treatment)
  NRS is suitable for the assessment of current pain severity as perceived by the participant using a 0-10 points scale. A score of 10 corresponds to the worst pain.
Mean change in number and severity of falls assessed by the Falls Questionnaire (intra-group and between-groups comparisons) | T0 (baseline); T1 (end of the treatment - 8 weeks); T2 (3 months after the end of treatment)
  Falls Questionnaire is used for the assessment of the frequency and severity of falls.
  It provides information on the modality of falls and the number of falls in the last 12 months.
  A superior number of falls suggests a lower balance (no range of score).
Perception of satisfaction to the treatment assessed with a subjective satisfaction questionnaire- 5 point Likert scale | T1 (end of the treatment - 8 weeks)
  A 5 points Likert scale is useful to assess subjective satisfaction from 0 (minimum) to 5 (maximum)

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Fondazione Don Gnocchi Firenze, Florence, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gualerzi A, Picciolini S, Carlomagno C, Terenzi F, Ramat S, Sorbi S, Bedoni M. Raman profiling of circulating extracellular vesicles for the stratification of Parkinson's patients. Nanomedicine. 2019 Nov;22:102097. doi: 10.1016/j.nano.2019.102097. Epub 2019 Oct 21. PMID 31648040
- [Background] Erdfelder, E., Faul, F., & Buchner, A. (1996). GPOWER: A general power analysis program. Behavior research methods, instruments, & computers, 28(1), 1-11.
- [Background] Ganesan M, Sathyaprabha TN, Gupta A, Pal PK. Effect of partial weight-supported treadmill gait training on balance in patients with Parkinson disease. PM R. 2014 Jan;6(1):22-33. doi: 10.1016/j.pmrj.2013.08.604. Epub 2013 Sep 8. PMID 24021298
- [Background] Tinetti ME. Performance-oriented assessment of mobility problems in elderly patients. J Am Geriatr Soc. 1986 Feb;34(2):119-26. doi: 10.1111/j.1532-5415.1986.tb05480.x. No abstract available. PMID 3944402
- [Background] Goetz CG, Tilley BC, Shaftman SR, Stebbins GT, Fahn S, Martinez-Martin P, Poewe W, Sampaio C, Stern MB, Dodel R, Dubois B, Holloway R, Jankovic J, Kulisevsky J, Lang AE, Lees A, Leurgans S, LeWitt PA, Nyenhuis D, Olanow CW, Rascol O, Schrag A, Teresi JA, van Hilten JJ, LaPelle N; Movement Disorder Society UPDRS Revision Task Force. Movement Disorder Society-sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS): scale presentation and clinimetric testing results. Mov Disord. 2008 Nov 15;23(15):2129-70. doi: 10.1002/mds.22340. PMID 19025984
- [Background] Tambasco N, Simoni S, Eusebi P, Ripandelli F, Brahimi E, Sacchini E, Nigro P, Marsili E, Calabresi P. The validation of an Italian version of the Freezing of Gait Questionnaire. Neurol Sci. 2015 May;36(5):759-64. doi: 10.1007/s10072-014-2037-5. Epub 2014 Dec 17. PMID 25515786
- [Background] Downie WW, Leatham PA, Rhind VM, Wright V, Branco JA, Anderson JA. Studies with pain rating scales. Ann Rheum Dis. 1978 Aug;37(4):378-81. doi: 10.1136/ard.37.4.378. PMID 686873
- [Background] Podsiadlo D, Richardson S. The timed "Up & Go": a test of basic functional mobility for frail elderly persons. J Am Geriatr Soc. 1991 Feb;39(2):142-8. doi: 10.1111/j.1532-5415.1991.tb01616.x. PMID 1991946
- [Background] Keus SH, Nieuwboer A, Bloem BR, Borm GF, Munneke M. Clinimetric analyses of the Modified Parkinson Activity Scale. Parkinsonism Relat Disord. 2009 May;15(4):263-9. doi: 10.1016/j.parkreldis.2008.06.003. Epub 2008 Aug 8. PMID 18691929
- [Background] Galeoto G, Colalelli F, Massai P, Berardi A, Tofani M, Pierantozzi M, Servadio A, Fabbrini A, Fabbrini G. Quality of life in Parkinson's disease: Italian validation of the Parkinson's Disease Questionnaire (PDQ-39-IT). Neurol Sci. 2018 Nov;39(11):1903-1909. doi: 10.1007/s10072-018-3524-x. Epub 2018 Aug 7. PMID 30088166
- [Background] Ruggiero C, Mariani T, Gugliotta R, Gasperini B, Patacchini F, Nguyen HN, Zampi E, Serra R, Dell'Aquila G, Cirinei E, Cenni S, Lattanzio F, Cherubini A. Validation of the Italian version of the falls efficacy scale international (FES-I) and the short FES-I in community-dwelling older persons. Arch Gerontol Geriatr. 2009;49 Suppl 1:211-9. doi: 10.1016/j.archger.2009.09.031. PMID 19836635
- [Background] Molino-Lova R, Sofi F, Pasquini G, Gori A, Vannetti F, Abbate R, Gensini GF, Macchi C; Mugello Study Working Group. The Mugello study, a survey of nonagenarians living in Tuscany: design, methods and participants' general characteristics. Eur J Intern Med. 2013 Dec;24(8):745-9. doi: 10.1016/j.ejim.2013.09.008. Epub 2013 Oct 11. PMID 24125724
- [Background] Ghisi M at al 2006, Beck Depression Inventory - II (BDI-II) Manuale. Firenze: O.S. Organizzazioni Speciali
- [Background] Santangelo G, Barone P, Abbruzzese G, Ferini-Strambi L, Antonini A; IRIS Study Group. Validation of the Italian version of Parkinson's disease-cognitive rating scale (PD-CRS). Neurol Sci. 2014 Apr;35(4):537-44. doi: 10.1007/s10072-013-1538-y. Epub 2013 Sep 25. PMID 24221858
- [Background] Giovagnoli AR, Del Pesce M, Mascheroni S, Simoncelli M, Laiacona M, Capitani E. Trail making test: normative values from 287 normal adult controls. Ital J Neurol Sci. 1996 Aug;17(4):305-9. doi: 10.1007/BF01997792. PMID 8915764
- [Background] Nocentini U, Giordano A, Di Vincenzo S, Panella M, Pasqualetti P. The Symbol Digit Modalities Test - Oral version: Italian normative data. Funct Neurol. 2006 Apr-Jun;21(2):93-6. PMID 16796824
- [Background] Aiello EN, Gramegna C, Esposito A, Gazzaniga V, Zago S, Difonzo T, Maddaluno O, Appollonio I, Bolognini N. The Montreal Cognitive Assessment (MoCA): updated norms and psychometric insights into adaptive testing from healthy individuals in Northern Italy. Aging Clin Exp Res. 2022 Feb;34(2):375-382. doi: 10.1007/s40520-021-01943-7. Epub 2021 Jul 27. PMID 34313961
- [Background] Chen ZY, Yan HJ, Qi L, Zhen QX, Liu C, Wang P, Liu YH, Wang RD, Liu YJ, Fang JP, Su Y, Yan XY, Liu AX, Xi J, Fang B. C-Gait for Detecting Freezing of Gait in the Early to Middle Stages of Parkinson's Disease: A Model Prediction Study. Front Hum Neurosci. 2021 Mar 22;15:621977. doi: 10.3389/fnhum.2021.621977. eCollection 2021. PMID 33828470
- [Background] Steffen T, Seney M. Test-retest reliability and minimal detectable change on balance and ambulation tests, the 36-item short-form health survey, and the unified Parkinson disease rating scale in people with parkinsonism. Phys Ther. 2008 Jun;88(6):733-46. doi: 10.2522/ptj.20070214. Epub 2008 Mar 20. Erratum In: Phys Ther. 2010 Mar;90(3):462. PMID 18356292
- [Background] Siciliano M, Chiorri C, Passaniti C, Sant'Elia V, Trojano L, Santangelo G. Comparison of alternate and original forms of the Montreal Cognitive Assessment (MoCA): an Italian normative study. Neurol Sci. 2019 Apr;40(4):691-702. doi: 10.1007/s10072-019-3700-7. Epub 2019 Jan 14. PMID 30637545
- [Background] Santangelo G, Lagravinese G, Battini V, Chiorri C, Siciliano M, Abbruzzese G, Vitale C, Barone P. The Parkinson's Disease-Cognitive Rating Scale (PD-CRS): normative values from 268 healthy Italian individuals. Neurol Sci. 2017 May;38(5):845-853. doi: 10.1007/s10072-017-2844-6. Epub 2017 Feb 21. PMID 28224328
- [Background] Wang Y, Gao L, Yan H, Jin Z, Fang J, Qi L, Zhen Q, Liu C, Wang P, Liu Y, Wang R, Liu Y, Su Y, Liu A, Fang B. Efficacy of C-Mill gait training for improving walking adaptability in early and middle stages of Parkinson's disease. Gait Posture. 2022 Jan;91:79-85. doi: 10.1016/j.gaitpost.2021.10.010. Epub 2021 Oct 11. PMID 34656008
- See also: gait parameters derived from Optogait assessment — http://www.optogait.com/Gait-Phases